CLINICAL TRIAL: NCT04108637
Title: Penicillin Allergy Status And Its Effect On Antibiotic Prescribing, Patient Outcomes, and Antimicrobial Resistance
Brief Title: Allergy Antibiotics And Microbial Resistance
Acronym: ALABAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Jonathan Sandoe, Associate Clinical Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: V14.0 16Nov2023
Record Dates: First submitted 2019-03-05; First posted 2019-09-30 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Infection
Keywords: penicillin; allergy; antimicrobial; resistance
MeSH Terms: conditions — Infections; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Multicentre, two parallel-arm, open label, individually randomised pragmatic trial with a nested-pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- penicillin allergy assessment pathway (Experimental): Those in the PAAP intervention arm will complete stage 2&3 of the PAAP pathway:
  * Stage-2 assessed for skin testing (ST) and ST done or straight to stage 3
  * Stage-3 oral challenge test (OCT) All completing PAAP will receive a letter from the immunology clinic giving the results of the test. Also, patients who have tested negative will receive the "Post-test Intervention Booklet" and "Patient Intervention Card" Materials.
  Additionally, all participants in the PAAP arm will be called by the trial team at days 4-6 and 28-30 post testing to collect safety data. During the call at days 28-30 patients will complete the patient questionnaire on allergy beliefs.
  Practices will be informed of the test result and instructed to update the participant's electronic health records accordingly.
  Interventions: Procedure: penicillin allergy assessment pathway
- Control Arm (No Intervention): The usual care arm receive no intervention but will be followed up as per intervention arm with monitoring of any symptoms following an antibiotic prescription.

INTERVENTIONS:
Procedure: penicillin allergy assessment pathway — Summary of penicillin allergy assessment pathway :
  Stage-1 PAAP in Primary Care - Clinical History. Screening, questionnaire and antimicrobial history will be undertaken in primary care Stage-2 Skin Test(ST) in hospital clinic (this may not be needed for all participants) Stage 3 Oral Challenge Test (OCT) in hospital clinic Testing will involve half a day in clinic and then a three-day post clinic course of oral antimicrobial therapy, without a reaction
  Other Names: PAAP
  Arms: penicillin allergy assessment pathway

SUMMARY:
ALBAMA study is designed to find out if the effects of Penicillin allergy assessment pathway (PAAP) intervention is on penicillin prescribing

DETAILED DESCRIPTION:
* Antibiotics are important medicines for fighting infections caused by bacteria. Their widespread use has caused a worrying rise in antibiotic resistant bacteria, which are bacteria that are harder to control or kill with antibiotics. Patients with infections caused by antibiotic resistant bacteria are often ill for longer and have an increased risk of serious harm, including death. The spread of resistant bacteria can be slowed down by using antibiotics more carefully. Penicillins are an important group of antibiotics that are recommended treatment for many infections. Doctors will avoid prescribing penicillin for their patients who have a "penicillin allergy label" in their health records. These patients are usually prescribed different types of antibiotics for their infections. There is concern that these non-penicillin antibiotics may not work as well as penicillins, may cause more side-effects (including killing more of the body's "helpful" bacteria), and may be more expensive.
* About 9 out of 10 people who have a record of penicillin-allergy are found to be not truly allergic to penicillin when thoroughly tested. This means they could safely take penicillins. The aim of ALABAMA is to find out if people with a penicillin-allergy record in their GP health records really do have an allergy by carrying out specialist testing, and to see if it is possible to reduce the number of patients wrongly labelled as penicillin allergic. The investigators will find out if this results in better use of antibiotics and fewer days of symptoms, when patients are prescribed antibiotics for infection.
* The investigators are recruiting up to 140 GP practices in Yorkshire and Humber and the South West Peninsula to help with this research, and plans to include up to 1060 people.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above
* Current penicillin allergy (or sensitivity) record of any kind in their electronic health record
* Receipt of either: penicillin, cephalosporin, tetracycline, quinolone or macrolide class antibiotic or fosfomycin, nitrofurantoin, trimethoprim, clindamycin in the previous 12 months

N.B.1 Patients who have been formally tested for penicillin allergy in the past and been found not to be penicillin allergic but still have a medical record indicating a penicillin allergy, are eligible for the trial.

Exclusion Criteria:

* Life expectancy estimated <1 year by GP

  * Unable to attend immunology clinic
  * Unsuitable for entry into testing pathway because:

    * Allergy history consistent with anaphylaxis to penicillin
    * History of toxic epidermal necrolysis, Stevens-Johnson syndrome, Drug reaction with eosinophilia and systemic symptoms (DRESS) or any severe rash which blistered or needed hospital treatment, and acute generalised exanthematous pustulosis precipitated by a penicillin
    * Has been formally tested for penicillin allergy in the past and been found to be penicillin allergic
    * History of brittle/severe asthma or has had a course of steroids in the past 3 months for asthma or unstable coronary artery disease, or dermographism or other severe/poorly controlled skin conditions
    * Considered unsuitable for trial participation by the GP e.g. because of chaotic lifestyle
  * Pregnant
  * Breastfeeding mothers
  * Taking beta blocker medication, and unable to temporarily withhold these on the day of penicillin allergy testing
  * Currently taking (or recently taken) systemic steroids and unable to stop these for 10 days pretesting.
  * Currently taking antihistamines and unable to temporarily withhold these for 72 hours pre-testing

GPs may also want to exclude vulnerable patients who are deemed to be unsuitable to participate for other reasons such as, but not limited to, terminal illness, reliability, mental illness, learning difficulties, anxiety, and other family circumstances.

N.B.1 Patients that are currently taking medicines with antihistamine properties that cannot be temporarily withheld, or patients with isolated dermographism, may still be eligible to participate but will need to be discussed with the research team prior to consent.

N.B.2 Pregnancy and breastfeeding exclusion criteria are only applicable at screening (due to potential risks of PAT); these patients would not need to be withdrawn if in follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Penicillin prescribing | Measured at up to 12 month post-randomisation
  The proportion of participants who receive prescriptions for a penicillin when attending for predefined conditions where a penicillin is the first-line recommended antibiotic

SECONDARY OUTCOMES:
Treatment "response failure" | Measured after first antibiotic prescription, which can occur any time during the follow-up period for patients(Up to 12 months post randomisation)
  Treatment "response failure" will be defined as: Re-presentation with worsening or non-resolving symptoms following treatment with an antibiotic up to 28 days after initial antibiotic prescription (including re-prescription of antibiotic within 28 days of an index prescription) for predefined conditions (TPP/notes review), over the year subsequent to randomisation. This will be compared between groups
Symptom duration | Measured up to 12 month post-randomisation
  Duration of symptoms (in days) rated 'moderately bad' or worse by patients, after initiation of antibiotic treatment
Total antibiotic prescribing | Measured up to 12 month post-randomisation
  Count of total antibiotic use (measured as total number of days therapy and as average daily quantity (ADQ) antibiotics. Total number of penicillin and each non-penicillin antibiotic prescriptions (measured as total number of days therapy and ADQ)
Hospital admissions | Measured up to 12 month post-randomisation
  Count of total number of hospital admissions
Length of hospital stays | Measured up to 12 month post-randomisation
  Count of total length of hospital stays
Mortality rates | Measured up to 12 month post-randomisation
  Mortality rates compared between intervention arms
Meticillin-resistant Staphylococcus aureus (MRSA) infection/ colonisation | Measured up to 12 month post-randomisation
  Total number of patients with MRSA infection/colonisation compared between intervention arms
Clostridium difficile infection | Measured up to 12 month post-randomisation
  Number of patients with Clostridium difficile infection
(Process evaluation) To explore patient and clinician experiences of trial procedures. | Within 12 months of practice recruitment of a proportion of tested patients
  GP and patient interviews
To measure changes in clinician and patient behaviour change regarding prescribing and consuming penicillin following a negative test result. | Within 12 months of practice recruitment of a proportion of tested patients
  Change in self-reported behaviour by clinicians and patients.
To measure the influences on clinician and patient behaviour change regarding prescribing and consuming penicillin following a negative test result. | Within 12 months of practice recruitment of a proportion of tested patients
  influences on behaviour by clinicians and patients.
Cost effectiveness for the PAAP intervention compared to usual care | Collated for period: randomisation to up to 12 months of randomisation
  Measurement of quality adjusted life years in each arm
De-labelling | check performed at 3 and 12 months
  The proportion of ALABAMA participants whose labels were removed and remain removed from the medical eHR

OTHER OUTCOMES:
AEs and SAEs reported | Measured at up to 12 month post-randomisation
  A descriptive analysis will be performed looking at the safety (number of AEs and SAEs) of de-labelling in the intervention group
Effects of PAAP on all outcomes for follow up past 12 months | Measured at the end of the study
  Descriptive analysis using data captured in the notes review CRF

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sandoe, Dr, Study Chair — University of Leeds
Locations (1):
- NIHR CRN: Yorkshire and Humber, York, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed S, Fielding J, Porter CE, Armitage KF, Wanat M, Bates C, Engonidou L, West RM, Yu LM, Galal U, Howard P, Butler CC, Savic S, Boards J, Tonkin-Crine S, Parry J, Pavitt SA, Sandoe JT; ALABAMA research team. Utilising primary care electronic health records to deliver the ALABAMA randomised controlled trial of penicillin allergy assessment. Trials. 2024 Oct 3;25(1):653. doi: 10.1186/s13063-024-08506-x. PMID 39363246
- [Derived] Wanat M, Santillo M, Galal U, Davoudianfar M, Bongard E, Savic S, Savic L, Porter C, Fielding J, Butler CC, Pavitt S, Sandoe J, Tonkin-Crine S; ALABAMA team. Mixed-methods evaluation of a behavioural intervention package to identify and amend incorrect penicillin allergy records in UK general practice. BMJ Open. 2022 Jun 3;12(6):e057471. doi: 10.1136/bmjopen-2021-057471. PMID 36691248

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04108637/SAP_000.pdf